CLINICAL TRIAL: NCT04630964
Title: The Effect of Psilocybin on MDD Symptom Severity and Synaptic Density - A Single Dose Randomized, Double Blind, Placebo- Controlled Phase 2 Positron Emission Tomography Study
Brief Title: The Effect of Psilocybin on MDD Symptom Severity and Synaptic Density
Acronym: PSIPET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Section for Affective Disorders; Northern Stockholm Psychiatry (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-002790-94
Record Dates: First submitted 2020-11-12; First posted 2020-11-16 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Psilocybin; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psilocybin (Experimental): 25 mg Single Oral Dose
  Interventions: Drug: Psilocybin
- placebo (Active Comparator): 100 mg Single Oral Dose
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: Psilocybin — psilocybin 25 mg Single Oral Dose
  Arms: psilocybin
Drug: Niacin — niacin 100mg Single Oral Dose
  Arms: placebo

SUMMARY:
PROTOCOL SYNOPSIS Title The effect of psilocybin on Major depressive disorder (MDD) symptom severity and synaptic density - a single dose randomized, double blind, placebo-controlled phase 2b positron emission tomography study Study Code PSIPET Name of Sponsor SLSO Organisationsnr: 232100-0016 Sponsor representative: Andreas Carlborg Norra Stockholms Psykiatri Vårdvägen 3 112 19 Stockholm Sweden Medical Monitor Inspira Medical AB Phase of Study Phase 2b Sample Size 30 randomized Name of Investigational Product (IP) Psilocybin, 3-[2-(dimethylamino)ethyl]-1H-indol-4-yl] dihydrogen phosphate Name of Active Placebo Niacin EudraCT 2020-002790-94 Description of IP and Active Placebo PSIPET Protocol 5 200821 Page 14 Study Intervention Name: Psilocybin (active drug product) Niacin (active placebo product) Dosage formulation: One active capsule contains 25 mg of psilocybin One active placebo capsule contains 100 mg of niacin Capsule: Size 2 hydroxypropyl methylcellulose (HPMC), opaque Size 2 HPMC, opaque Unit dose strength: 25 mg 100 mg Route of Administration: Oral (solid dose) Oral (solid dose) Dosing instructions: One capsule administered with water One capsule administered with water Packaging and Labeling: Study Intervention will be provided in a high-density polyethylene (HDPE) bottle. Each bottle will contain one capsule (psilocybin or niacin) and will be labeled as required per Swedish requirement for blinded study.

DETAILED DESCRIPTION:
Study Description and Overview Thirty participants (males and females) ages 20 to 65 inclusive, who, at Screening, meet ICD-10 criteria for major depressive disorder (MDD), have a current depressive episode of at least 30-day duration, have a Screening Montgomery-Asberg Depression Rating Scale (MADRS) total score >= 22 and meet all other inclusion/exclusion criteria will be randomized with a 1-to-1 allocation under double-blind conditions to receive a single 25 mg oral dose of psilocybin or a single 100 mg oral dose of niacin. Niacin will serve as an active placebo control that provides an acute physiological response (flushing) that is intended to aid in blinding of intervention allocation. All randomized participants will be included in the Full Analysis Set (FAS) population used in analyzing primary and secondary study endpoints. Only participants who meet depressive symptom severity criteria at web screening (MADRS self-rating (MADRS-S) score > =19) and who do not show an unacceptably large degree of symptom improvement between the web screening and in-person screening (indexed by change in MADRS-S (improvement) 30% (MADRS representing web screening will be approximated to MADRS-S + 3) will be eligible for randomization. This is to minimize the risk for spontaneous remission before dosing. Participants deemed eligible following successful completion of all screening assessments including a structural Magnetic Resonance Imaging (MRI) examination will be determined as eligible. Eligible participants at Baseline will submit cerebrospinal fluid (CSF), submit blood samples, be examined with positron emission tomography (PET) and the radioligand [11C]UCB-J and receive one preparation session (see further below) to be eligible for randomization on Dosing (Day 0) to receive either psilocybin or niacin active-placebo. They will complete follow-up visits, including outcome measures assessments, on study Day 1, 8, 15, 42 and 365 (within corresponding visit windows). At day 15 the sampling of CSF, blood and [11C]UCB-J PET will be repeated. PSIPET Protocol 5 200821 Page 15 After day 42, all participants will be given follow-up visits at Norra Stockholms Psykiatri for up to one year after dosing, to study dedicated physicians or nurses at a frequency determined by the health care professional. If needed to reach/stay in remission, the participants will be provided antidepressant treatment in accordance with the regional guidelines for antidepressant treatment (https://psykiatristod.se/regionala-vardprogram/ depression). At least monthly the participants will be asked to provide on-line symptom rating data (via 1177.se). At the 365-day visit, symptoms will be evaluated using MADRS, Clinical Global Impression Improvement (CGI-I) and Severity (CGI-S) scales. After completing the study (one year or withdrawal), participants will be subject to standard care, including referral in accordance with regional guidelines. The study outcome measures will be used to assess depressive symptoms, clinical global functioning, functional disability, anxiety symptoms and health-related quality of life. Safety outcome measures will be collected at all assessment time points from the time of consent through the end of study. To enhance participant safety, the current study proposes to test psilocybin within a "set and setting" (SaS) protocol similar to the protocol that has been used in all modern studies of psilocybin in both diseased and normal healthy populations. The SaS protocol for this study includes: 1) a preparation with session Facilitators (licensed psychologists) prior to dosing; 2) administration of study medications in an aesthetically neutral room under the supervision of two Facilitators who are present throughout the session (with the exception of short, temporary allowances for facilitator breaks; e.g. bathroom breaks); and 3) three post-dose integration sessions during which participants are encouraged to discuss their intervention experience with the Facilitators. To evaluate the Facilitators' adherence to the study manual, and the role of Facilitators' and participants' in-session behaviors for treatment outcome, all five sessions in the trial with Facilitators present will be recorded. The SaS will be identical for those randomized to psilocybin or niacin active placebo. Study Duration The planned maximum study duration for each participant will be approximately one year, with variation primarily dependent on the length of the screening period, the number of days between baseline and dosing, and the visit windows provided for each post-dose assessment. For each participant, the study will be divided into two phases: Phase A or treatment phase (day 0 to and including day 42), and phase B or follow-up phase (day 43 -365). The primary objective of this study is to evaluate the efficacy of a single 25 mg oral dose of psilocybin for major depressive disorder (MDD) compared to an active placebo (niacin) in otherwise medically-healthy participants between the ages of 20 and 65, assessed as the difference between groups in changes in depressive symptoms. Primary Outcome Measure Change in blinded rater MADRS total score from Baseline to Day 8.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to be randomized in this protocol are those who meet all of the following criteria:

1. Are 20 to 65 years old at the time of written informed consent at the In-Person Screening visit
2. Are able to read, speak, and understand Swedish
3. Are able and willing to adhere to study requirements, including attending all study visits, preparatory and follow-up sessions, and completing all study evaluations
4. Are able to swallow capsules
5. Women of childbearing potential (WOCBP) must agree to practice an effective means of birth control throughout the duration of the study, from Screening through the Day 42 assessment
6. Meet ICD-10 criteria for a diagnosis of remitting major depressive disorder and are currently experiencing a major depressive episode of

   1. at least a 30-day duration at the time of the Screening
   2. less than 5 years at time of Screening
7. Have sustained moderate-severe depression symptoms at Screening and Baseline, as defined by a Screening MADRS total score ≥ 22 and ≤30% and ≤7 point improvement (i.e. decrease) in MADRS total score from web-screening to screening visit (assuming 3 points on item 1 at web screening).

9. Have an identified support person

a. Agree to be driven/accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing

-

Exclusion Criteria:

Individuals not eligible to be randomized in this protocol are those who meet any of the following criteria:

1. Women who are pregnant, as indicated by a positive urine pregnancy test at Screening or Baseline. Women who intend to become pregnant during the study or who are currently nursing.
2. Current depressive episode lasting >5 years

2. Unwilling or unable to discontinue formal psychotherapy 3. Ongoing antidepressant drug treatment 4. Have previously during the current episode received the following non-medication treatments:

a. deep brain stimulation (DBS) b. vagus nerve stimulation (VNS) 5. Currently receiving electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) 6. Unable or unwilling to discontinue any current medications that are known uridine diphosphate (UDP) or glucuronosyltransferase (UGT) enzyme modulators (eg valproate)

* Note: Any prohibited agents must have been stopped at least 5x the elimination half-life of the specific drug at the time of Baseline. See Appendix A for a full list of prohibited medications.

  7. Report psychedelic substances use ever
* Note: Psychedelic substances include psilocybin, Lysergic acid diethylamide (LSD), mescaline (and natural products containing mescaline including peyote and San Pedro cactus), N,N-Dimethyltryptamine (DMT), natural products containing DMT including ayahuasca and 5-Methoxy-N,N-dimethyltryptamine (5-MeO-DMT), ibogaine, 2C compounds, 3,4-methylenedioxy- methamphetamine (MDMA), methylone or other psychedelics.

  8. Have the following cardiovascular conditions:

  a. coronary artery disease, congenital long QT syndrome (prior diagnosis), cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction (prior diagnosis); b. tachycardia (defined as heart rate > 100 beats per minute); c. a clinically significant Screening ECG abnormality (e.g., atrial fibrillation); oNote: A QTcF interval > 450 milliseconds is considered a clinically significant ECG abnormality d. artificial heart valve; or e. any other significant current or history of cardiovascular condition, based on the clinical judgment of study physician, that would make a participant unsuitable for the study 9. At Screening or Baseline have elevated blood pressure as defined as:

  a. Screening blood pressure SBP >135 mmHg or DBP > 85 mmHg on three separate readings; or b. Baseline blood pressure SBP >140 mmHg or DBP > 90 mmHg on three separate readings 10. Have a history of stroke or Transient Ischemic Attack (TIA) 11. Have moderate to severe hepatic impairment, as indexed by a Child-Pugh score ≥ 7 12. Have epilepsy 13. Have insulin-dependent diabetes
* Note: Participants who are taking oral hypoglycemic agent and have a history of hypoglycemia requiring medical intervention will be excluded 14. Are unable or unwilling to adhere to the following medication requirements:

  1. Agree to suspend sildenafil (Viagra®), tadalafil, or similar medications at least 72 hours prior to dosing
  2. If taking any supplement containing >20 mg of niacin, agrees to suspend use for the duration of the study 15. Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Cannabis, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP), and Tetrahydrocannabinol (THC). Exceptions are made for prescribed Benzodiazepines (stable dose for sleep or anxiety).
* Note: Benzodiazepine medications for sleep and non-benzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for at least 6 weeks prior to Screening, as determined during review of concomitant medications
* Note: Participants using cannabis, including legal cannabis, for any purposes will be excluded
* Note: Participants who are taking prescription maintenance methadone or buprenorphine naloxone will be excluded
* Note: Prescription opiates must have been stopped at least 5x the elimination half- life of the specific drug at the time of inclusion, as confirmed with a negative urine drug screen.

  16. Nicotine dependence that would disallow an individual to be nicotine free for the 7-10 hours during the dosing period 17. Meet ICD-10 criteria for schizophrenia spectrum or other psychotic disorders, including MDD with psychotic features (except substance/medication-induced or due to another medical condition), or Bipolar I Disorder, Bipolar II Disorder and bipolar disorder NOS.
* Note: Participants with any lifetime diagnosis of schizophrenia spectrum or other psychotic disorders will be excluded 18. Meet ICD-10 criteria for antisocial personality disorder 19. Meet ICD-10 criteria for a moderate or severe alcohol or drug use disorder (excluding caffeine)
* Note: Participants with a diagnosis of alcohol or drug use disorder within the past 12 months will be excluded 20. Have presence of any psychiatric condition or symptom judged by the PI (or designee) to be a more significant clinical problem than MDD for the participant.

  21. Have a first-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I Disorder 22. Have a psychiatric condition judged to be incompatible with establishment of rapport with the Facilitators or safe exposure to psilocybin 23. Report the following suicidal ideation or suicidal thoughts defined as:

  a. Have a score of ≥ 5 on Item 10 (suicidal thoughts) of the central-rater or computer administered MADRS at Screening or Baseline; or b. Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior at any time prior to randomization 24. Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior 25. Have any physical or psychological symptom, medication or other relevant finding at Screening or Baseline, based on the clinical judgment of clinical/medical study personnel, that would make a participant unsuitable for the study.

  26. Have an allergy or intolerance to any of the materials contained in either drug product 27. Have Hepatitis B, C or HIV 28. Have one or more pathological blood test results as defined in 5.6.3 (as determined by a study physician; with the exception of CRP).

  29. Have peptic ulcer (ICD 10 K25 or K26)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale (MADRS) | 8 days
  Change in blind rater MADRS total score. MADRS range: 0-60. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
[11C]UCB-J | 7 to 1 day before dosing to 15 +/-7 days after dosing.
  Change in UCB-J binding as measured using PET

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Stockholm Spychiatry Clinic, Stockholm, Sweden